CLINICAL TRIAL: NCT05651178
Title: A Early Phase 1 Clinical Trial to Evaluate the Safety and Efficacy of Human CD19-CD22 Targeted T Cells Injection for Subjects with Central Nervous System Involvement of Refractory/Relapsed B Cell Malignancies
Brief Title: Human CD19-CD22 Targeted T Cells Injection for Refractory/Relapsed Central Nervous System Leukemia/Lymphoma Patients
Status: Recruiting | Phase: Early Phase 1 | Type: Interventional
Sponsor: Hrain Biotechnology Co., Ltd. (Industry)
Collaborators: Second Affiliated Hospital of Nanchang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HRAIN02-CNSL01
Record Dates: First submitted 2022-12-02; First posted 2022-12-14 (Actual); Last update posted 2025-01-07 (Actual); Status verified 2024-12

CONDITIONS: Central Nervous System Lymphoma
Keywords: CD19-CD22; CAR-T; Central nervous system leukemia/lymphoma; Refractory/Relapsed
MeSH Terms: conditions — Lymphoma; Recurrence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Human CD19-CD22 Targeted T Cells Injection (Experimental): Intravenous administration: 1.0×10^6 CAR+T cells/kg, 3.0×10^6 CAR+T cells/kg, 5.0×10^6 CAR+T cells/kg. Intrathecal administration: The initial dose is set at 1 × 10⁶ CAR+cells per patient. The decision to escalate the intrathecal dose and frequency is made based on the condition of the subjects.
  Interventions: Drug: Human CD19-CD22 Targeted T Cells Injection

INTERVENTIONS:
Drug: Human CD19-CD22 Targeted T Cells Injection — Autologous genetically modified anti-CD19/CD22 CAR transduced T cells
  Other Names: CD19-CD22 CAR-T

SUMMARY:
This study is a open-label, dose-escalation trial to explore the safety, tolerability and pharmacokinetic/pharmacodynamics characteristics of Human CD19-CD22 Targeted T Cells by intravenous and intrathecal administration, and to preliminarily observe the efficacy of the trial drug in patients with central nervous system involvement of refractory/relapsed B cell malignancies.

DETAILED DESCRIPTION:
Subjects with refractory/relapsed central nervous system involvement of B cell malignancies can participate if all eligibility criteria are met. Tests required to determine eligibility including disease assessments, a physical exam, Electrocardiograph, Computed tomography (CT) / Magnetic Resonance Imaging (MRI) / Positron Emission Tomography (PET), Cerebrospinal fluid exam and blood draws. Subjects will receive preconditioning chemotherapy prior to the infusion of Human CD19-CD22 Targeted T Cells Injection. After the infusion, subjects will be followed for adverse events, pharmacokinetic/pharmacodynamics characteristics, efficacy of Human CD19-CD22 Targeted T Cells Injection. Study procedures may be performed while hospitalized.

ELIGIBILITY:
Inclusion Criteria:Subjects must meet all of the following criteria to be enrolled:

* B cell malignancies patients with CD19 or CD22 positive, or CD19 and CD22 positive，include B cell acute lymphoblastic leukemia relapsed with central nervous system invasion and refractory/relapsed B cell lymphoma of central nervous system;
* 18 to 70 years old (including cut-off value), Male and female;
* Expected survival > 12 weeks;
* ECOG score 0-2;
* Definitive diagnosed as central nervous system of B cell malignancies by Cerebrospinal fluid and/or MRI, PET/CT or other imaging examinations;
* The venous access required for collection can be established and leukapheresis can be carried according to the judgement of investigators;
* Liver, kidney and cardiopulmonary functions meet the following requirements:

  1. The detection value of Creatinine within the normal range;
  2. Left ventricular ejection fraction > 50%;
  3. Baseline oxygen saturation > 92%;
  4. Total bilirubin ≤ 2×ULN;
  5. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5×ULN;
* Able to understand and sign the Informed Consent Document.

Exclusion Criteria:Any one of the following conditions cannot be selected as a subject:

* Malignant tumors other than B cell malignancies within 5 years prior to screening, in addition to adequately treated cervical carcinoma in situ, basal cell or squamous cell skin cancer, localized prostate cancer after radical resection, ductal carcinoma in situ after radical resection and thyroid cancer after radical resection;
* Subjects with positive Hepatitis B surface antigen (HBsAg) or Hepatitis B core antibody (HBcAb) and peripheral blood hepatitis B virus (HBV) DNA titer detection higher than or equal to the lower limit of detection; hepatitis C virus (HCV) antibody positive and peripheral blood HCV RNA positive; human immunodeficiency virus (HIV) antibody positive; syphilis detection positive;
* Any instability of systemic disease, including but not limited to unstable angina, cerebrovascular accident, or transient cerebral ischemic (within 6 months prior to screening), myocardial infarction (within 6 months prior to screening), congestive heart failure (New York heart association (NYHA) classification ≥ III), need drug therapy of severe arrhythmia, liver, kidney, or metabolic disease;
* Active or uncontrollable infection requiring systemic therapy within 14 days prior to enrollment;
* Pregnant or lactating woman, and female subject who plans to have a pregnancy within 1 year after cell transfusion, or male subject whose partner plans to have a pregnancy within 1 year after cell transfusion;
* Received CAR-T treatment or other gene therapies before enrollment;
* Subjects who are receiving systemic steroid treatment and requiring long-term systemic steroid treatment during the treatment as determined by the investigator before screening (except inhalation or topical use); And subjects treated with systemic steroids (except inhalation or topical use) within 72h prior to cell infusion;
* The investigators consider other conditions unsuitable for enrollment.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2022-08-12 (Actual); Primary Completion 2024-11-30 (Actual); Study Completion 2025-08-31 (Estimated)

PRIMARY OUTCOMES:
Dose limited toxicity (DLT) | 28 days post infusion
  Safety Indicators
The occurrence rate of adverse events grade ≥ 3 assessed by NCI-CTCAE 5.0 | 28 days post infusion
  Safety Indicators

SECONDARY OUTCOMES:
Pharmacokinetics parameters - the highest concentration of Human CD19-CD22 Targeted T Cells amplified in peripheral blood after reinfusion | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - the time to reach the highest concentration of Human CD19-CD22 Targeted T Cells amplified in peripheral blood after reinfusion | 2 years post infusion
  Effectiveness Metrics
Pharmacokinetics parameters - the 28-day area under the curve of Human CD19-CD22 Targeted T Cells amplified in peripheral blood after reinfusion | 2 years post infusion
  Effectiveness Metrics
The rate of CAR-T cells in cerebrospinal fluid | 2 years post infusion
  Effectiveness Metrics
The duration of CAR-T cells in cerebrospinal fluid | 2 years post infusion
  Effectiveness Metrics
Pharmacodynamics characteristics - the detection values of IL-6, IFN-γ, IL-15 cytokines in peripheral blood | 2 years post infusion
  Effectiveness Metrics
Overall response rate (ORR) at 3 months after administration | 3 months post infusion
  Effectiveness Metrics
Duration of remission (DOR) after administration | 2 years post infusion
  Effectiveness Metrics
Overall Survival (OS) after administration | 2 years post infusion
  Effectiveness Metrics

CONTACTS AND LOCATIONS:
Overall Officials: Qingming Wang, M.D., Principal Investigator — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Affiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No